CLINICAL TRIAL: NCT01533571
Title: Immediate Implant Placement After Tooth Extraction in the Esthetic Zone: Extraction Socket Morphology-Guided Treatment Modalities and Esthetic Outcome
Brief Title: Immediate Implant Placement in the Esthetic Zone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Lithuanian University of Health Sciences (Other)
Collaborators: Hacettepe University (Other); Universidad de Granada (Other); University of Michigan (Other)
Responsible Party: Principal Investigator, Povilas Daugela, Principal Investigator, Lithuanian University of Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Juodzbalys
Record Dates: First submitted 2012-02-07; First posted 2012-02-15 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Unspecified Atrophy of Edentulous Alveolar Ridge
Keywords: Guided Bone Regeneration; Dental Implant; Alveolar Ridge Augmentation; Socket graft
MeSH Terms: interventions — cerabone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate implant + xenogenic graft (Active Comparator): Treatment with immediate implant and GBR using xenogenic bone graft material
  Interventions: Procedure: Immediate implant placement with simultaneous bone grafting
- Immediate implant + allogenic graft (Active Comparator): Treatment with immediate implant and GBR using allogenic bone graft material.
  Interventions: Procedure: Immediate implant placement with simultaneous bone grafting

INTERVENTIONS:
Procedure: Immediate implant placement with simultaneous bone grafting — * Flapless surgery is used for surgical implant installation.
  * Implant is placed in the cingulum position of adjacent teeth incisal edge.
  * After placement of optimal implant the remaining gap between the implant and the surrounding bony walls should be at least 2 mm or should be need for GBR of buccal plate outside the socket.
  * Two types of bone graft materials will be applied for two groups of patients: Group I - natural bovine bone grafting material + resorbable natural soft tissue membrane; Group II - processed human allograft + resorbable natural soft tissue membrane .
  Crown can be fixed on abutment if there is initial stability under 35 Ncm insertion torque. If insertion torque will be less, crown should be bond to neighboring teeth using composite material.
  Other Names: Cerabone; Jason membrane; Maxgarft; Straumann Bone level implant

SUMMARY:
This study aims to examine dimensional alveolar ridge alterations and prevent buccal plate resorption and soft tissue recession following immediate implant placement in extraction sockets in the maxillary esthetic zone using different socket morphology-guided treatment modalities.

Expected results of the study are:

* To have found the optimal materials and GBR procedures modalities for buccal plate resorption degree reduction;
* Soft tissue recession and best esthetic result achievement. There will be possibilities to study socket morphology influence on final esthetic result achievement.

DETAILED DESCRIPTION:
Aim of the study: to examine dimensional alveolar ridge alterations and prevent buccal plate resorption and soft tissue recession following immediate implant placement in extraction sockets in the maxillary esthetic zone using different socket morphology-guided treatment modalities.

Objectives:

* To evaluate extraction socket buccal plate resorption rate among patients groups with immediate implant placement simultaneously with guided bone regeneration (GBR) methods using different types of bone graft materials.
* To evaluate esthetic outcome using Complex Esthetic Index (CEI) (Appendix 3) and correlate this to the initial buccal plate thickness and soft tissue biotype assessed during immediate implant placement simultaneously with GBR.
* To recommend the most appropriate method for prevention of buccal plate resorption, soft tissue recession and esthetic result achievement following immediate implant placement in extraction sockets in the maxillary esthetic zone.

Methods

Patients sampling:

* Selection of patients with sufficient extraction sockets for immediate dental implant installation with guided bone regeneration (GBR) procedure.
* Assessment of the extraction socket should be done using classification of extraction socket based upon soft and hard tissue components before the treatment (Appendix 2).

Result analysis

Size of the research:

Sixty patients referred to an oral implantologist in Kaunas, Vilnius, Granada, Ankara cities that need immediate implants in the esthetic zone. There will be 2 groups of patients:

1. Group I patients (n = 30) treated with immediate implant and GBR using xenogenic bone graft material;
2. Group II patients (n = 30) treated with immediate implant and GBR using allogenic bone graft material.

Expected result:

After the study, we hope to have found the optimal materials and GBR procedures modalities for buccal plate resorption degree reduction, soft tissue recession and best esthetic result achievement. There will be possibilities to study socket morphology influence on final esthetic result achievement.

Funds:

Private sponsorship, companies sponsorship (Straumann and Botiss Dental). Detailed Protocol

After patient selection there will be few steps in present study (you can press Ctrl-Enter and go directly to the selected step):

Step 1. Clinical examination and documentation Conventional clinical examination will be done. Orthopantomograph and standardized periapical radiograph will be registered for every patient. Informed consent should be signed. Additionally an acrylic stent will be fabricated for each subject. This stent will be fixed on the incisal edges of the adjacent teeth taking into consideration planned acrylic temporary tooth space. The stent will provide three buccal/lingual pairs of consistent measurement points for each implant site located 4, 7, and 10 mm from the summit of the alveolar soft tissue. One aperture 1 will be above soft tissue margin. We should insert into aperture 1 cylinder with constant length until it contact most prominent implant transfer part. Then assistant should add acrylic or composite resin into aperture and fix cylinder strongly into template by this way. Thus we will have constant distance from point 1 to the implant collar (5 or 6mm according to the need).

Step 2. Tooth extraction Following local anesthesia, the teeth should be gently extracted, using 15c blades, periotomes, elevators and forceps, minimizing any fractures of the socket walls. Sites are thoroughly degranulated for proper visualization and clinical assessment of the socket morphology.

Step 3. Socket assessments and classification Below is an overview of extraction socket classification (Appendix 2 and Figure 1). As stated before, this classification is derived from present soft and hard tissue variables.

1. Soft tissue contour variations;
2. Vertical soft tissue deficiency;
3. The keratinized gingival (KG) width on the mid-buccal side of the socket;
4. Mesial and distal papillae appearance
5. Gingival tissue biotype;
6. Soft tissue quality;
7. The height of alveolar process;
8. Available bone beyond the apex of extraction socket;
9. Extraction socket labial plate vertical position;
10. Extraction socket facial bone thickness;
11. Presence of extraction socket bone lesions;
12. Intra-dental bone peak height (interproximal bone height);
13. The mesio-distal (M-D) distance between adjacent;
14. Palatal angulation.

All linear measurements will be performed to the closest 1 mm with the use of a periodontal probe. All measurements will be done by two surgeons and mean will be calculated.

Step 4. Dental implant placement. All implants should be placed in the optimal three dimensional position. Dental implant should be placed in the cingulum position (in line with adjacent teeth) and planned implant tooth incisal edge position should be in line with adjacent teeth incisal edge. In this ideal position, the implant collar should be 2 mm below the cementoenamel junction of the adjacent teeth apicocoronally or 3-4 mm bellow planned soft tissue margin, and at least 1.5 mm away from adjacent teeth mesiodistally.

After placement of optimal dental implant the remaining gap between the implant and the surrounding bony walls should be at least 2 mm or should be need for GBR of buccal plate outside the socket.

Step 5. Implant position and alveolar bone assessment:

1. Bone in front to the implant width;
2. Bucco-lingual ridge width;
3. Vertical residual gap;
4. Implant apico-coronal position. Step 6. The remaining defects augmentation based on the proposed scheme. Flapless surgery will be applied consequently GBR application place will be inside the socket. The remaining defects and dehiscences after implant placement will be filled up, using two types of bone graft materials: Group I - natural bovine bone grafting material + resorbable natural soft tissue membrane and Group II - processed human allograft + resorbable natural soft tissue membrane. In future we will call Group II control group. Resorbable membrane should be condensed on bone graft without pressure and fixed by provisional crown. Conventional medicament treatment including Chlorhexidine 0.2% oral rinses twice daily for 2 weeks will be applied.

Step 7. The provisional crown fixation. Individualized provisional acrylic crown will be fabricated before operation and will be adapted and fixed on temporary abutment after implant insertion if there is initial implant stability under 35 Ncm insertion torque. The provisional crown will be cemented with temporary cement. If the implant fails to achieve initial stability under 35 Ncm insertion torque, the provisional acrylic crown would be bonded to the neighboring teeth. In all cases, the provisional crowns are excluded from occlusion. After 6 months, the provisional restorations will be replaced by a permanent cemented or screw-retained zirconia crown.

Step 8. Final prosthetic treatment After 6 months, the provisional restorations will be replaced by a permanent cemented zirconia crown fixed on zirconia abutment. Patients follow up: Patients will be rechecked two times: 6 months and 1 year after implant treatment.

Step 10. Complex Esthetic Index (CEI) for anterior maxillary implant supported restorations This complex esthetic index is composed of three components: the soft tissue index (S), predictive index (P) and implant supported restoration index (R) (Appendix 1).

Appendix 1. Clinical documentation sequence:

1. Preoperative picture of mouth area of patient, including smile line
2. Clinical preoperative picture of defect area (approximately 4 teeth in picture)
3. Preoperative orthopantomography and periapical X-ray
4. Extraction of the tooth
5. Socket measurements with caliper and probe
6. Operation area ready for implantation
7. Implant placement
8. Bone substitute application
9. Resorbable membrane application
10. Clinical situation right after surgery with the provisional crown
11. Clinical situation postoperative 1 week (if available)
12. Clinical situation postoperative 6 months without provisional crown (incisal edges and frontal view projections)
13. Clinical situation postoperative 6 months with permanent crown (incisal edges and frontal view projections)
14. Follow-up after 6 months periapical X-ray
15. Alveolar process measurements with caliper and probe
16. Clinical situation postoperative 1 year after treatment (incisal edges and frontal view projections)
17. Follow-up after 1 year periapical X-ray
18. Alveolar process measurements with caliper and probe

Appendix 2. Extraction socket soft and hard tissue assessments and socket types questionnaire Observer:_________________ Assessment series No □

Date:

Cause for tooth loss:

Patients name and family name:

Gender: Male □ Female □

Tooth No: 15 14 13 12 11 21 22 23 24 25

Soft and hard tissues assessment

Extraction socket types: Adequate Compromised Deficient

Soft tissue Quantity

Soft tissue contour variations No □ <2 mm □ ≥2 mm □

Soft tissue vertical deficiency (probe) No □ 1 to 2 mm □ >2 mm □

Keratinized gingival width (probe) >2 mm □ 1 to 2 mm □ <1 mm □

Mesial and distal papillae appearance (Nordland & Tarnow) I □ II □ III □

Soft tissue color, consistency, and contour Pink, firm and smooth □ Slightly red, soft sponge and uneven contour □ Red/Bluish, red, soft oedematous and boggy or craterlike soft tissue appearance □

Biotype of gingival tissue (probe) Thick □ Moderate □ Thin □ 2.0 mm □ ≥1.0 to <2.0 mm □ <1.0 mm □

Hard tissue Height of alveolar process (orthopantomograph) >10 mm □ >8 to ≤10 mm □ ≤8 mm □

Available bone beyond the apex of extraction socket (orthopantomograph) ≥4 mm □ ≥3 to <4 mm □ <3 mm □

Extraction socket labial plate vertical position; (probe) ≤3 mm □ >3 to <7 mm □ ≥7 mm □

Extraction socket facial bone thickness (caliper) ≥2 mm □ ≥1 to <2 mm □ <1 mm □

Presence of socket bone lesions No □ Yes □ Yes □

Mesial and distal intra-dental bone peak height (periapical X-ray) 3 to 4 mm □ ≥1 to <3 mm □ <1 mm □

Mesio-distal distance between adjacent teeth (probe) ≥7 mm □ >5 to <7 mm □ ≤5 mm □

The need for palatal angulation (diagnostic wax-up) <5° □ 5-30° □ >30° □

Extraction socket type:

Appendix 3. Complex Esthetic Index (CEI) questionnaire Observer:_________________ Assessment series No □

Date:

Patients name and family name:

Index and parameters Rating and evaluation grades of parameters variations Adequate 20% Compromised 10% Deficient 0%

S index

1. Soft tissue contour variations (probe) No □ <2mm □ ≥2mm □
2. Soft tissue vertical deficiency (probe) No □ 1 to 2 mm □ >2 mm □
3. Soft tissue color and texture variations No □ Moderate □ Obvious □
4. Mesial papillae appearance Complete fill □ Partial fill □ None □
5. Distal papillae appearance Complete fill □ Partial fill □ None □

S index general rating and evaluation grade 100% 60-90% <50%

P index

1. Mesial interproximal bone height (periapical X-ray) <5 mm □ 5 to 7 mm □ >7 mm □
2. Distal interproximal bone height (periapical X-ray) <5 mm □ 5 to 7 mm □ >7 mm □
3. Gingival tissue biotype (probe) >2 mm □ 1 to 2 mm □ <1 mm □ 4

Implant apico-coronal position (probe) 1.5 to 3 mm □ >3 to5 mm □ >5 mm □ 5

Horizontal contour deficiency (probe) No □ 1 to 3 mm □ >3 mm □

P index general rating and evaluation grade 100% 60-90% <50%

R index

1. Color and translucency No □ Moderate □ Obvious □
2. Labial convexity in the abutment/implant junction No □ <1 mm □ <2 mm □
3. Implant/crown incisal edge position No □ ±1mm □ ±2 mm □
4. Crown width/length ratio <0.85 □ 0.85 to 1.0 □ >1.0 □
5. Surface roughness and ridges No □ Moderate □ Obvious □

R index general rating and evaluation grade 100% 60-90% <50%

Gender: Male □ Female □

Tooth No: 15 14 13 12 11 21 22 23 24 25

Complex Esthetic Index: S¬____% P____% R____%.

ELIGIBILITY:
Inclusion Criteria:

* General health satisfactory
* Single-tooth replacement in the maxillary anterior segments
* Extraction socket Type I and Type II (Juodzbalys et al.)
* Non-adjacent implant sites and prosthetic restorations
* Patient will not wear any kind of removable prosthesis over the treatment area;
* Availability of complete clinical records.

Exclusion Criteria:

* Uncontrolled diabetes
* Immunodeficiency diseases
* Heavy smokers (more than 10 cigarettes a day)
* Untreated periodontal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-04 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Complex Esthetic Index (CEI) | One year
  CEI will be evaluated by two calibrated observers and mean will be calculated. Complex esthetic index is composed of three components: the soft tissue index (S), predictive index (P) and implant supported restoration index (R).

CONTACTS AND LOCATIONS:
Overall Officials: Gintaras Juodzbalys, Professor, Study Chair — Lithuanian University of Health Sciences (Lithuania); Hom-Lay Wang, Professor, Study Chair — University of Michigan; Pablo Galindo-Moreno, Professor, Principal Investigator — University of Granada (Spain); Tolga F Tozum, Professor, Principal Investigator — Hacettepe University (Turkey); Povilas Daugela, Dr., Principal Investigator — Lithuanian University of Health Sciences (Lithuania); Algirdas Puisys, Dr., Principal Investigator — Lithuanian University of Health Sciences (Lithuania)
Locations (4):
- University of Michigan, Ann Arbor, Michigan, United States
- Lithuanian University of Health Sciences, Kaunas, Lithuania
- University of Granada, Granada, Spain
- Hacettepe University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Juodzbalys G, Wang HL. Socket morphology-based treatment for implant esthetics: a pilot study. Int J Oral Maxillofac Implants. 2010 Sep-Oct;25(5):970-8. PMID 20862411
- [Background] Juodzbalys G, Wang HL. Esthetic index for anterior maxillary implant-supported restorations. J Periodontol. 2010 Jan;81(1):34-42. doi: 10.1902/jop.2009.090385. PMID 20059415
- [Background] Juodzbalys G, Sakavicius D, Wang HL. Classification of extraction sockets based upon soft and hard tissue components. J Periodontol. 2008 Mar;79(3):413-24. doi: 10.1902/jop.2008.070397. PMID 18315423
- [Background] Juodzbalys G, Bojarskas S, Kubilius R, Wang HL. Using the support immersion endoscope for socket assessment. J Periodontol. 2008 Jan;79(1):64-71. doi: 10.1902/jop.2008.070253. PMID 18166094
- [Background] Juodzbalys G, Wang HL. Soft and hard tissue assessment of immediate implant placement: a case series. Clin Oral Implants Res. 2007 Apr;18(2):237-43. doi: 10.1111/j.1600-0501.2006.01312.x. PMID 17348889
- [Background] Nordland WP, Tarnow DP. A classification system for loss of papillary height. J Periodontol. 1998 Oct;69(10):1124-6. doi: 10.1902/jop.1998.69.10.1124. PMID 9802711
- See also: Journal of Oral & Maxillofacial Research (JOMR) — http://www.ejomr.org